CLINICAL TRIAL: NCT04920955
Title: Evaluation of a Novel Blood Multi-marker Test for the Detection of Colorectal Cancer Relapse
Brief Title: Relapse Markers for Colorectal Cancer
Acronym: RELMA-C
Status: Completed | Type: Observational
Sponsor: Novigenix SA (Other)
Responsible Party: Sponsor
Other Study IDs: S64663
Record Dates: First submitted 2021-06-02; First posted 2021-06-10 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral whole blood and Plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- G1, CRC Relapse: Patients with an actual relapse of CRC, within 5 years from primary surgery. A single blood sample is collected at relapse diagnosis.
- G2, CRC Disease-free: Patients previously diagnosed with CRC and declared disease-free for at least 36 months but less than 5 years. A single blood sample is collected at standard monitoring visit.
- G3, CRC Disease-free (longitudinal): Patients declared disease-free for at least 3 months but less than 18 months. Longitudinal blood samples will be collected during standard monitoring visits up to relapse, or for a maximum of 4 time points.
- G4, Primary CRC (longitudinal): Patients with an actual diagnosis of CRC who are eligible for a treatment with curative intent. Blood samples will be collected pre and post-surgery (~6 weeks) and, eventually, at relapse.

SUMMARY:
This is an observational case-control study which enroll metastatic and non-metastatic colorectal cancer (CRC) patients. The objective of this study is to evaluate a novel blood multi-marker test for the detection of relapse in colorectal cancer patients. This test is based on whole-blood transcriptomic signatures and circulating tumor methylated DNA markers. The patients will be enrolled into 4 study groups, two cross-sectional and two longitudinal groups, to follow up patients up to 36 months from primary tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age at time of informed consent.
* Subject has signed the informed consent form (ICF) and is able to understand the information provided in it.
* At least a blood sample is collected per subject according to the sample collection protocol.
* Patients enrolled in local prospective protocols, in which samples have been collected according the study procedures may be included.
* Group 1: patients with a radiologically and, whenever is possible, histologically confirmed relapse (local or distant) of colorectal cancer within 5 years from primary surgery. Metachronous primary tumors are not considered as relapse and should be excluded.
* Group 2: Patients declared disease-free for at least 36 months but less than 5 years, as confirmed by radiological examination.
* Group 3: Patients with a stage III-IV colorectal cancer with a curative treatment and disease-free for at least 3 months but less than 18 months.
* Group 4: Histologically and radiologically confirmed diagnosis of stage I, II, III or IV colorectal adenocarcinoma, eligible for a treatment with curative intent.

Exclusion Criteria:

* Personal history of cancer (non-hematologic) other than CRC in complete remission for less than 5 years.
* Personal history of hematologic cancer.
* A blood transfusion within 6 weeks prior to inclusion into the study.
* Transplant with regular intake of immunosuppressants.
* Pregnant woman (self-declaration).
* Conditions or comorbidities that would preclude the compliance with the planned surveillance program or with the protocol as judged by the Investigator.
* Previous inclusion in the RELMA-C study and/or re-inclusion in a different study group.
* Group 1: Any treatment for CRC relapse prior to blood collection.
* Group 2: Patient is disease-free for less than 36 months or more than 5 years.
* Group 3: Patient is disease-free for less than 3 months or more than 18 months
* Group 3: Stage IV patients with detectable residual disease after primary treatment.
* Group 4: Any cancer treatment prior to blood collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll CRC patients into 4 study groups. G1: patients with an actual diagnosis of CRC relapse. G2: patients declared disease-free for at least 36 months but less than 5 years.
  G3: stage III-IV CRC patients who underwent a curative treatment and are disease-free after primary treatment for more than 3 but less than 18 months.
  G4: patients diagnosed with primary CRC without any cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity for relapse detection | Relapse occurring within 5 years from primary curative intervention
  Sensitivity of the test for detection of CRC relapse using radiological imaging as the reference diagnostic method
Specificity for relapse detection | 36 months disease-free
  Specificity of the test for detection of CRC relapse using radiological imaging as the reference diagnostic method

SECONDARY OUTCOMES:
Concordance analyses | 24 months
  Concordance analyses between the multi-marker and Carcinoembryonic Antigen (CEA) test for all patients and time points
Test positivity | 24 months
  Estimation of the multi-marker test positivity for all patients and time points
Coefficient of variation of the biomarkers | 6 weeks
  Intra- and inter-individual coefficient of variation of the biomarkers, pre- and post-surgery and during surveillance up to relapse
Sensitivity for CRC detection | up to 1 day prior to tumor resection
  Sensitivity of the test for detection of primary CRC

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ciarloni, Study Director — Novigenix SA; Sabine Tejpar, Principal Investigator — UZ Leuven
Locations (1):
- Department of Gastroenterology, Digestive Oncology Unit, Leuven, Belgium